CLINICAL TRIAL: NCT04739761
Title: An Open-Label, Multinational, Multicenter, Phase 3b/4 Study of Trastuzumab Deruxtecan in Patients With or Without Baseline Brain Metastasis With Previously Treated Advanced/Metastatic HER2-Positive Breast Cancer (DESTINY-Breast12)
Brief Title: A Study of T-DXd in Participants With or Without Brain Metastasis Who Have Previously Treated Advanced or Metastatic HER2 Positive Breast Cancer
Acronym: DESTINY-B12
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9673C00007; 2024-510588-53-00 (Registry Identifier: CTIS (EU)); 2020-005048-46 (EudraCT Number)
Record Dates: First submitted 2021-01-20; First posted 2021-02-05 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Trastuzumab deruxtecan; Human epidermal growth factor receptor 2 Positive Breast Cancer; Brain Metastasis
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trastuzumab Deruxtecan (Experimental): Participants with or without BM at baseline will receive intravenous (IV) T-DXd, 5.4 mg/kg, every 3 weeks (21-day cycle) until Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) defined radiological progression outside central nervous system, unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met.
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Participants will receive T-DXd administered using an IV bag containing 5% (w/v) dextrose injection infusion solution.
  Other Names: fam-trastuzumab deruxtecan-nxki

SUMMARY:
This is open-label, multicenter, international study, assessing the efficacy and safety of Trastuzumab deruxtecan (T-DXd) in participants with or without brain metastasis (BMs), with previously-treated advanced/metastatic HER2-positive breast cancer whose disease has progressed on prior anti-HER2-based regimens and who received no more than 2 lines/regimens of therapy in the metastatic setting (excluding tucatinib).

DETAILED DESCRIPTION:
Approximately 500 eligible participants will be enrolled into 1 of 2 cohorts (250 participants in each cohort) according to the presence or absence of BMs at baseline. Cohort 1 will include participants without BM at baseline and Cohort 2 will consist of participants with BM at baseline.

After study intervention discontinuation, all participants will undergo an end-of-treatment visit (within 7 days of discontinuation) and will be followed up for safety assessments 40 (+ up to 7) days after the discontinuation of all study intervention.

All participants will be followed up for survival status and duration of treatment on subsequent therapies after intervention discontinuation every 3 months (± 14 days) from the date of the safety follow-up until death, withdrawal of consent, or the end of the study, as per defined in the protocol.

ELIGIBILITY:
Inclusion:

* Participants should have pathologically documented breast cancer that is: unresectable/advanced or metastatic; confirmed HER2-positive status expression as determined according to American Society of Clinical Oncology/College of American Pathologists guidelines
* Participant must have either: no evidence of BM, or untreated BM on screening contrast brain magnetic resonance imaging/ computed tomography (MRI/CT) scan, not needing immediate local therapy or previously-treated stable or progressing BM
* Participants with BMs must be neurologically stable
* For participants requiring radiotherapy due to BMs, there should be an adequate washout period before day of first dosing:
* ≥ 7 days since stereotactic radiosurgery or gamma knife
* ≥ 21 days since whole brain radiotherapy
* Eastern Cooperative Oncology Group performance status 0-1
* Previous breast cancer treatment: radiologic or objective evidence of disease progression on or after HER2 targeted therapies and no more than 2 lines/regimens of therapy in the metastatic setting
* Participant with the following measurable: at least 1 lesion that can be accurately measured at baseline as ≥ 10 mm in the longest diameter with CT or MRI and is suitable for accurate repeated measurements; or following Non-measurable diseases: Non-measurable, bone-only disease that can be assessed by CT or MRI or X-Ray. Lytic or mixed lytic bone lesions that can be assessed by CT or MRI or X-ray in the absence of measurable disease as defined above is acceptable; Participants with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible; and Non-measurable CNS disease (Cohort 2 only)
* Adequate organ and bone marrow function within 14 days before the day of first dosing as defined in the protocol
* Left ventricular ejection fraction ≥ 50% within 28 days before enrollment
* Negative pregnancy test (serum) for women of childbearing potential

Exclusion Criteria

* Known or suspected leptomeningeal disease
* Prior exposure to tucatinib treatment
* Refractory nausea and vomiting, chronic gastrointestinal disease, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of T-DXd
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study intervention and of low potential risk for recurrence
* Based on screening contrast brain MRI/CT scan, participants must not have any of the following: any untreated brain lesions > 2.0 cm in size; ongoing use of systemic corticosteroids for control of symptoms of BMs; any brain lesion thought to require immediate local therapy; have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to BMs not withstanding CNS-directed therapy
* Has spinal cord compression
* Known active hepatitis B or C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1. Participants with past or resolved hepatitis B virus infection are eligible, if negative for hepatitis B surface antigen and positive for anti-hepatitis B core antigen
* Participants positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of T-DXd
* Participants with a medical history of myocardial infarction within 6 months before screening, symptomatic congestive heart failure (New York Heart Association Class II to IV)
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Lung-specific intercurrent clinically significant illnesses and any autoimmune, connective tissue or inflammatory disorders
* Prior exposure, without adequate treatment washout period before the day of first dosing, to chloroquine/hydroxychloroquine: < 14 days
* Anticancer chemotherapy: immunotherapy (non-antibody-based therapy), retinoid therapy, hormonal therapy: < 3 weeks
* < 6 weeks for nitrosoureas or mitomycin
* Antibody-based anticancer therapy: < 4 weeks
* Any concurrent anticancer treatment. Concurrent use of hormonal therapy for noncancer- related conditions is allowed
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline
* Palliative radiotherapy with a limited field of radiation within 2 weeks or with wide field of radiation, radiation to the chest, or to more than 30% of the bone marrow within 4 weeks before the first dose of study intervention
* Participants with prior exposure to immunosuppressive medication within 14 days prior to first study dose
* Participants with a known hypersensitivity to study intervention or any of the excipients of the product or other monoclonal antibodies

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2026-05-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, MD, PhD, Principal Investigator — Head, Breast Center, Ludwig-Maximilians-University of Munich Department of Obstetrics and Gynecology Marchioninistr. 15, 81377 Munich, Germany; Nancy U. Lin, MD, Principal Investigator — Associate Chief, Division of Breast Oncology, Susan F. Smith Center for Women's Cancers Director, Metastatic Breast Cancer Program, Dana-Farber Cancer Institute, 450 Brookline Avenue, Boston, MA 02215
Locations (73):
- United States (2):
  - Research Site, Boston, Massachusetts
  - Research Site, Durham, North Carolina
- Australia (6):
  - Research Site, Adelaide
  - Research Site, Auchenflower
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, St Leonards
  - Research Site, Subiaco
- Belgium (4):
  - Research Site, Anderlecht
  - Research Site, Bruges
  - Research Site, Leuven
  - Research Site, Liège
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
- Denmark (3):
  - Research Site, Copenhagen
  - Research Site, Herlev
  - Research Site, Odense C
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
- Germany (12):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Münster
  - Research Site, Tübingen
- Ireland (2):
  - Research Site, Cork
  - Research Site, Dublin
- Italy (7):
  - Research Site, Ancona
  - Research Site, Bergamo
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Prato
- Japan (5):
  - Research Site, Isehara
  - Research Site, Kawasaki-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Yokohama
- Netherlands (2):
  - Research Site, Maastricht
  - Research Site, The Hague
- Norway (2):
  - Research Site, Bergen
  - Research Site, Oslo
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Opole
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Santiago de Compostela-Coruña
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Uppsala
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Bellinzona
  - Research Site, Lausanne
  - Research Site, Lucerne
- Research Site, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Harbeck N, Ciruelos E, Jerusalem G, Muller V, Niikura N, Viale G, Bartsch R, Kurzeder C, Higgins MJ, Connolly RM, Baron-Hay S, Gion M, Guarneri V, Bianchini G, Wildiers H, Escriva-de-Romani S, Prahladan M, Bridge H, Kuptsova-Clarkson N, Scotto N, Verma S, Lin NU; DESTINY-Breast12 study group. Trastuzumab deruxtecan in HER2-positive advanced breast cancer with or without brain metastases: a phase 3b/4 trial. Nat Med. 2024 Dec;30(12):3717-3727. doi: 10.1038/s41591-024-03261-7. Epub 2024 Sep 13. PMID 39271844
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673C00007&attachmentIdentifier=fc591080-ce57-4a38-a7fb-4f0d73d8a6b2&fileName=AZ_D9673C00007_(PXL_254020)_Statistical_analysis_plan_Redacted_26_July_2024_Final_Approved_pdfa.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673C00007&attachmentIdentifier=30ed5660-a312-4e15-9fc7-fa666cae8a51&fileName=AZ_D9673C00007_(PXL_254020)_Protocol_Amendment_#2_07Jun2022_Redacted_Final_to_Sponsor_pdfa.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673C00007&attachmentIdentifier=03f0e826-3d81-4840-873f-e1ab50845c99&fileName=AZ_D9673C00007_(PXL_254020)_CSR_Synopsis_Final_Sponsor_approved_Redacted_pfda.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 22 June 2021 (First participant in) and the analyses presented in this results form are based on a final data cut-off of 08 February 2024 and final database lock of 22 April 2024.
Pre-assignment Details: Participants meeting eligibility criteria predefined in protocol were enrolled in the study. Assessments were to be performed as per the schedule of the assessments. However, 2 participants were in early withdrawal status since they completed enrollment but never received any treatment.
Groups:
- Cohort 1: Trastuzumab Deruxtecan (T-DXd): Participants without brain metastasis at baseline received T-DXd in Cohort 1 of the study.
- Cohort 2: Trastuzumab Deruxtecan (T-DXd): Participants with brain metastasis at baseline received T-DXd in Cohort 2 of the study.
Period: Overall Study
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Started | 241 | 263
Completed (A participant was considered to have completed the study when participant either died or withdrew from study after completing the safety follow-up visit or the survival follow-up visit.) | 30 | 34
Not Completed | 211 | 229
Not completed — Participant ongoing study at data cutoff date of 08Feb24 | 167 | 189
Not completed — By complete response from the participant | 1 | 0
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 13 | 13
Not completed — Participant reports worsening of the general critical condition and will not continue | 0 | 1
Not completed — Participant is in poor health and will not come to the study site | 0 | 1
Not completed — Progression confirmed in magnetic resonance imaging | 0 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Participant decision | 1 | 0
Not completed — Sub investigator decision approved by medical monitor | 1 | 0
Not completed — Participant immediately started next line of treatment | 1 | 0
Not completed — Participant's decision because the treatment makes them anxious | 1 | 0
Not completed — Lack of clinical benefit | 1 | 0
Not completed — Disease progression | 5 | 5
Not completed — Withdrawal by Subject | 14 | 13
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd) | Total
Number analyzed (Participants) | 241 | 263 | 504
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (11.9) | 52.8 (11.2) | 53.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 263 | 504
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — For Single participant in a particular race, the data was not reported under specific race, rather customised option was used, and the data was reported as Other to maintain participant's confidentiality
  Participants
    Asian | 15 | 19 | 34
    Black or African American | 2 | 4 | 6
    White | 209 | 231 | 440
    Other | 13 | 6 | 19
    Not reported | 1 | 1 | 2
    Missing | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 20 | 15 | 35
  Not Hispanic or Latino | 219 | 245 | 464
  Missing | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Cohort 1 (Participants Without Brain Metastasis at Baseline)
Description: The ORR is defined as the percentage (%) of participants who have a confirmed complete response (CR) or confirmed partial response (PR), as determined by independent central review (ICR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Time Frame: From first dose (Day 1) to progression of disease (up to 2 years 7 months)
Population: The full analysis set (FAS) included all participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241
Percentage of participants | 62.7 [56.5 to 68.8]

2. Primary Outcome: Progression-free Survival (PFS) Rate at 12 Months in Cohort 2 (Participants With Brain Metastasis at Baseline)
Description: The PFS rate is the percentage of participants alive and free of disease progression at 12 months, estimated by the Kaplan-Meier method.
Time Frame: At 12 months
Population: The FAS set included all the participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 263
Percentage of participants | 61.6 [54.92 to 67.61]

3. Secondary Outcome: Survival Rate at 12 Months
Description: Survival rate is the percentage of participants alive at 12 months, estimated by the Kaplan-Meier method.
Time Frame: At 12 Months
Population: The FAS included all participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241 | 263
Percentage of Participants | 90.6 [85.97 to 93.80] | 90.3 [85.89 to 93.41]

4. Secondary Outcome: Objective Response Rate in Cohort 2 (Participants With Brain Metastasis at Baseline)
Description: The ORR is defined as the percentage of participants who have a confirmed CR or confirmed PR, as determined by ICR per RECIST 1.1.
Time Frame: From first dose (Day 1) to progression of disease (up to 2 years 7 months)
Population: The FAS included all the participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 263
Percentage of participants | 51.7 [45.7 to 57.8]

5. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 as assessed by ICR or death due to any cause.
Time Frame: From the date of first documented confirmed response until date of documented progression (up to 2 years 7 months)
Population: The FAS included all participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241 | 263
Months | NA [9.5 to NA] — In line with methods prespecified in the SAP, the median and 75th percentile were not calculable because <50% of participants had an event. | NA [8.1 to NA] — In line with methods prespecified in the SAP, the median and 75th percentile were not calculable because <50% of participants had an event.

6. Secondary Outcome: Time to Progression
Description: Time to progression by RECIST 1.1 per ICR is defined as the time from the date of the first dose of study intervention to the date of documented disease progression.
Time Frame: From first dose (Day 1) to progression of disease (up to 2 years 7 months)
Population: The FAS included all the participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241 | 263
Months | NA [NA to NA] — As pre-specified in SAP, median and 95% confidence interval (CI) were not calculable where less than 50% of participants had events. | NA [NA to NA] — As pre-specified in SAP, median and 95% CI were not calculable where less than 50% of participants had events.

7. Secondary Outcome: Duration of Treatment on Subsequent Lines of Therapy
Description: Duration of treatment on subsequent therapy is defined as the time from the date of first dose of a subsequent therapy until date of the last dose of that therapy.
Time Frame: From the date of first dose of a subsequent therapy until date of last dose of therapy (up to 2 years 7 months)
Population: The Full analysis set-subsequent therapy included all participants in FAS had RECIST progression, as assessed by investigator, during the study and received subsequent anti-cancer therapy. The "number analyzed" refers to the number of participants included in analysis in specific time points in each row.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 68 | 66
Months
  First subsequent line of therapy | 4.4 [3.3 to 6.3] | 6.5 [3.9 to 8.8]
  First completed subsequent line of therapy: number analyzed (Participants) | 41 | 33
  First completed subsequent line of therapy | 3.0 [2.1 to 3.5] | 3.0 [2.1 to 3.5]

8. Secondary Outcome: Second Progression-Free Survival Rate at 12 Months
Description: Second progression-free survival rate is the percentage of participants alive and free from a second progression on next-line treatment at 12 months, estimated by the Kaplan-Meier method. The second progression is defined as the earliest progression event subsequent to the first anti-cancer therapy after the initial progression.
Time Frame: At 12 Months
Population: The FAS included all the participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241 | 263
Percentage of Participants | 81.1 [74.85 to 85.92] | 83.1 [77.46 to 87.44]

9. Secondary Outcome: Incidence of New Symptomatic Central Nervous System (CNS) Metastasis During Treatment Without CNS Metastasis at Baseline (Cohort 1)
Description: The incidence rate is defined as proportion of participants with new symptomatic CNS metastases during treatment period in participants without symptomatic CNS metastasis at baseline.
Time Frame: From first dose (Day 1) to end of treatment (up to 2 years 7 months)
Population: The FAS included all the participants who were involved in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241
Proportion of participants | 0.017 [0.00452 to 0.04250]

10. Secondary Outcome: Time to Next Progression (CNS or Extracranial) or Death
Description: The time to next progression is defined as the time from the date of the first documented isolated CNS progression to the date of the next documented disease progression (CNS or extracranial) per RECIST 1.1 or death and has been summarized descriptively in participants who have developed isolated CNS progression, receive local therapy, and continue on protocol therapy.
Time Frame: From date of first documented isolated CNS progression to the date of the next documented disease progression (up to 2 years 7 months)
Population: The FAS for isolated CNS progression analyses included participants that received at least 1 dose of treatment who developed isolated CNS progression, per investigator assessment, received local therapy, and continued on protocol therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 2 | 18
Months | 3.7 [3.7 to NA] — As pre-specified in SAP, upper limit of 95% CI was not calculable where less than 50% of participants had events. | 0.2 [0.1 to 0.3]

11. Secondary Outcome: Site (CNS vs Extracranial vs Both) of Next Progression
Description: Site of next progression (CNS [CNS RECIST 1.1] or extracranial [systemic RECIST 1.1] in participants who developed isolated CNS progression, received local therapy, and continued on protocol therapy.
Time Frame: From the date of the first documented isolated CNS progression to the date of the next documented CNS disease progression (up to 2 years 7 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 2 | 18
Participants
  CNS | 0 | 6
  Extracranial | 0 | 2
  Both | 0 | 4

12. Secondary Outcome: Central Nervous System Progression-free Survival Rate at 12 Months in Participants With Brain Metastasis at Baseline (Cohort 2)
Description: Central nervous system progression free survival rate is the percentage of participants free from central nervous system progression at 12 months, estimated by the Kaplan-Meier method.
Time Frame: At 12 Months
Population: The FAS included all the participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 263
Percentage of Participants | 58.9 [51.93 to 65.30]

13. Secondary Outcome: Time to New CNS Lesions in Participants With Brain Metastasis at Baseline (Cohort 2)
Description: The time to new CNS lesions is defined as the time from the date of the first dose of study intervention to the date of documented new CNS lesions by RECIST 1.1 per ICR.
Time Frame: From first dose (Day 1) to the date of documented new CNS lesions (up to 2 years 7 months)
Population: The FAS included all participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 263
Months | NA [NA to NA] — As pre-specified in SAP, median and 95% CI were not calculable where less than 50% of participants had events.

14. Secondary Outcome: Central Nervous System Objective Response Rate in Participants With Brain Metastasis at Baseline by ICR (Cohort 2)
Description: The CNS ORR is defined as the percentage of participants with measurable brain metastasis at baseline who have a confirmed CR or confirmed PR of brain lesions, as determined by ICR per CNS RECIST 1.1.
Time Frame: From first dose (Day 1) until CNS progression of disease (up to 2 years 7 months)
Population: The FAS included all participants who were enrolled in the study and received at least 1 dose of treatment. Here, number of participants analyzed represents participants who had measurable CNS disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 138
Percentage of participants | 71.7 [64.2 to 79.3]

15. Secondary Outcome: Central Nervous System Duration of Response in Participants With Brain Metastasis at Baseline (Cohort 2)
Description: The CNS DoR is defined as the time from the date of first documented confirmed CNS response until date of documented CNS progression per CNS RECIST 1.1 as assessed by ICR or death due to any cause.
Time Frame: From date of first documented confirmed CNS response until CNS progression of disease (up to 2 years 7 months)
Population: The FAS included all participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 263
Months | NA [6.9 to NA] — In line with methods prespecified in the SAP, the median and 75th percentile were not calculable because <50% of participants had an event.

16. Secondary Outcome: Number of Participants With Best on Treatment Visit Response on the European Organization for the Research and Treatment of Cancer 30-Item Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a 30-item questionnaire for cancer assessment. Increased scores indicate improvement; decreased scores indicate deterioration. Physical function: ≥+9= improvement, ≤-10=deterioration, otherwise=no change; Role functioning: ≤-6=deterioration, otherwise=no change; Social functioning: ≥+8=improvement, ≤-7=deterioration, otherwise=no change; Cognitive functioning: ≥+ 5=improvement, ≤- 4=deterioration, otherwise=no change; Global Health Status: ≥+2=improvement, ≤-8=deterioration, otherwise=no change; Fatigue: ≥+8=improvement, ≤-8=deterioration, otherwise=no change; Nausea and vomiting: ≤-11=deterioration, otherwise=no change; Appetite loss: ≤-14=deterioration, otherwise=no change; rest of scales: ≥+10=improvement, ≤-10=deterioration, otherwise=no change. Best on treatment response is best response category (improvement, no change, and deterioration) achieved by participants between first dose and 47 days after last dose, and prior to starting any anticancer therapy.
Time Frame: Time from first dose up to 47 days after last dose, or prior to starting any subsequent therapy, or for up to 2 years 7 months, whichever occurred first
Population: The safety analysis set included all the participants who have received at least 1 dose of treatment. The "overall number of participants analyzed" represents only participants who were not missing baseline data. The "number analyzed" refers to the number of participants included in each row for each response category.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 207 | 224
Participants
  Appetite loss: Best on-treatment response: Deterioration | 15 | 9
  Appetite loss: Best on-treatment response: No change | 171 | 200
  Appetite loss: Best on-treatment response: No follow-up | 21 | 15
  Appetite loss: Best on-treatment response: Missing | 0 | 0
  Cognitive Functioning: Best on-treatment response: Deterioration: number analyzed (Participants) | 207 | 223
  Cognitive Functioning: Best on-treatment response: Deterioration | 16 | 12
  Cognitive Functioning: Best on-treatment response: Improvement: number analyzed (Participants) | 207 | 223
  Cognitive Functioning: Best on-treatment response: Improvement | 57 | 87
  Cognitive Functioning: Best on-treatment response: No change: number analyzed (Participants) | 207 | 223
  Cognitive Functioning: Best on-treatment response: No change | 116 | 107
  Cognitive Functioning: Best on-treatment response: No follow-up: number analyzed (Participants) | 207 | 223
  Cognitive Functioning: Best on-treatment response: No follow-up | 18 | 17
  Cognitive Functioning: Best on-treatment response: Missing: number analyzed (Participants) | 207 | 223
  Cognitive Functioning: Best on-treatment response: Missing | 0 | 0
  Constipation: Best on-treatment response: Deterioration | 18 | 13
  Constipation: Best on-treatment response: Improvement | 36 | 59
  Constipation: Best on-treatment response: No change | 134 | 139
  Constipation: Best on-treatment response: No follow-up | 19 | 13
  Constipation: Best on-treatment response: Missing | 0 | 0
  Diarrhoea: Best on-treatment response: Deterioration: number analyzed (Participants) | 207 | 223
  Diarrhoea: Best on-treatment response: Deterioration | 2 | 4
  Diarrhoea: Best on-treatment response: Improvement: number analyzed (Participants) | 207 | 223
  Diarrhoea: Best on-treatment response: Improvement | 32 | 28
  Diarrhoea: Best on-treatment response: No change: number analyzed (Participants) | 207 | 223
  Diarrhoea: Best on-treatment response: No change | 153 | 174
  Diarrhoea: Best on-treatment response: No follow-up: number analyzed (Participants) | 207 | 223
  Diarrhoea: Best on-treatment response: No follow-up | 20 | 17
  Diarrhoea: Best on-treatment response: Missing: number analyzed (Participants) | 207 | 223
  Diarrhoea: Best on-treatment response: Missing | 0 | 0
  Dyspnea: Best on-treatment response: Deterioration | 6 | 5
  Dyspnea: Best on-treatment response: Improvement | 48 | 49
  Dyspnea: Best on-treatment response: No change | 131 | 154
  Dyspnea: Cycle Best on-treatment response: No follow-up | 22 | 16
  Dyspnea: Best on-treatment response: Missing | 0 | 0
  Emotional Functioning: Best on-treatment response: Deterioration: number analyzed (Participants) | 207 | 223
  Emotional Functioning: Best on-treatment response: Deterioration | 4 | 7
  Emotional Functioning: Best on-treatment response: Improvement: number analyzed (Participants) | 207 | 223
  Emotional Functioning: Best on-treatment response: Improvement | 109 | 98
  Emotional Functioning: Best on-treatment response: No change: number analyzed (Participants) | 207 | 223
  Emotional Functioning: Best on-treatment response: No change | 77 | 103
  Emotional Functioning: Best on-treatment response: No follow-up: number analyzed (Participants) | 207 | 223
  Emotional Functioning: Best on-treatment response: No follow-up | 17 | 15
  Emotional Functioning: Best on-treatment response: Missing: number analyzed (Participants) | 207 | 223
  Emotional Functioning: Best on-treatment response: Missing | 0 | 0
  Fatigue: Best on-treatment response: Deterioration | 28 | 23
  Fatigue: Best on-treatment response: Improvement | 97 | 119
  Fatigue: Best on-treatment response: No change | 65 | 68
  Fatigue: Best on-treatment response: No follow-up | 17 | 14
  Fatigue: Best on-treatment response: Missing | 0 | 0
  Financial difficulties: Best on-treatment response: Deterioration: number analyzed (Participants) | 206 | 223
  Financial difficulties: Best on-treatment response: Deterioration | 7 | 9
  Financial difficulties: Best on-treatment response: Improvement: number analyzed (Participants) | 206 | 223
  Financial difficulties: Best on-treatment response: Improvement | 46 | 58
  Financial difficulties: Best on-treatment response: No change: number analyzed (Participants) | 206 | 223
  Financial difficulties: Best on-treatment response: No change | 135 | 140
  Financial difficulties: Best on-treatment response: No follow-up: number analyzed (Participants) | 206 | 223
  Financial difficulties: Best on-treatment response: No follow-up | 18 | 16
  Financial difficulties: Best on-treatment response: Missing: number analyzed (Participants) | 206 | 223
  Financial difficulties: Best on-treatment response: Missing | 0 | 0
  Global health status / QoL: Best on-treatment response: Deterioration: number analyzed (Participants) | 207 | 223
  Global health status / QoL: Best on-treatment response: Deterioration | 28 | 34
  Global health status / QoL: Best on-treatment response: Improvement: number analyzed (Participants) | 207 | 223
  Global health status / QoL: Best on-treatment response: Improvement | 86 | 111
  Global health status / QoL: Best on-treatment response: No change: number analyzed (Participants) | 207 | 223
  Global health status / QoL: Best on-treatment response: No change | 75 | 65
  Global health status / QoL: Best on-treatment response: No follow-up: number analyzed (Participants) | 207 | 223
  Global health status / QoL: Best on-treatment response: No follow-up | 18 | 13
  Global health status / QoL: Best on-treatment response: Missing: number analyzed (Participants) | 207 | 223
  Global health status / QoL: Best on-treatment response: Missing | 0 | 0
  Insomnia: Best on-treatment response: Deterioration | 8 | 7
  Insomnia: Best on-treatment response: Improvement | 87 | 103
  Insomnia: Best on-treatment response: No change | 92 | 98
  Insomnia: Best on-treatment response: No follow-up | 20 | 16
  Insomnia: Best on-treatment response: Missing | 0 | 0
  Nausea and vomiting: Best on-treatment response: Deterioration | 17 | 9
  Nausea and vomiting: Best on-treatment response: No change | 167 | 201
  Nausea and vomiting: Best on-treatment response: No follow-up | 23 | 14
  Nausea and vomiting: Best on-treatment response: Missing | 0 | 0
  Pain: Best on-treatment response: Deterioration | 4 | 8
  Pain: Best on-treatment response: Improvement | 91 | 115
  Pain: Best on-treatment response: No change | 94 | 89
  Pain: Best on-treatment response: No follow-up | 18 | 12
  Pain: Best on-treatment response: Missing | 0 | 0
  Physical Functioning: Best on-treatment response: Deterioration | 10 | 13
  Physical Functioning: Best on-treatment response: Improvement | 54 | 71
  Physical Functioning: Best on-treatment response: No change | 122 | 124
  Physical Functioning: Best on-treatment response: No follow-up | 21 | 16
  Physical Functioning: Best on-treatment response: Missing | 0 | 0
  Role Functioning: Best on-treatment response: Deterioration | 20 | 15
  Role Functioning: Best on-treatment response: No change | 167 | 197
  Role Functioning: Best on-treatment response: No follow-up | 20 | 12
  Role Functioning: Best on-treatment response: Missing | 0 | 0
  Social Functioning: Best on-treatment response: Deterioration: number analyzed (Participants) | 207 | 223
  Social Functioning: Best on-treatment response: Deterioration | 19 | 16
  Social Functioning: Best on-treatment response: Improvement: number analyzed (Participants) | 207 | 223
  Social Functioning: Best on-treatment response: Improvement | 81 | 109
  Social Functioning: Best on-treatment response: No change: number analyzed (Participants) | 207 | 223
  Social Functioning: Best on-treatment response: No change | 87 | 83
  Social Functioning: Best on-treatment response: No follow-up: number analyzed (Participants) | 207 | 223
  Social Functioning: Best on-treatment response: No follow-up | 20 | 15
  Social Functioning: Best on-treatment response: Missing: number analyzed (Participants) | 207 | 223
  Social Functioning: Best on-treatment response: Missing | 0 | 0

17. Secondary Outcome: Number of Participants With Neurologic Assessment in Neuro-Oncology Scale (NANO Scale)
Description: The NANO scale is a clinician-reported assessment of neurologic functioning in neuro-oncology participants. The instrument captures 9 domains (gait, strength, ataxia, sensation, visual fields, facial strength, language, level of consciousness, and behavior) and was developed to provide a simple, objective assessment of neurologic function that would be combined with radiographic assessment to provide an overall outcome assessment for neuro-oncology participants in clinical trials and in daily practice. The soring scale for Gait consists of score range 0-3, Strength consists of score range 0-2, ataxia (upper extremity) consists of scale range 0-2 and sensation as 0. Higher scores indicate worse neurologic function. The response categories reported are changes from first post-baseline score to worst on-treatment score at any point of treatment.
Time Frame: as for outcome 16
Population: The FAS included all the participants who were enrolled in the study and received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 236 | 254
Participants
  Neurologic response | 3 | 4
  Neurologic stability | 217 | 220
  Neurologic progression | 16 | 25
  Not assessed | 0 | 5
  Non-evaluable | 0 | 0

18. Secondary Outcome: Cognitive Functions Tests: Paired Associates Learning (PAL) First Attempt Memory Score (PALFAMS)
Description: The PAL is a computerized, self-completed cognitive test used to capture cognitive function, including attention, memory, and executive function. This gamified test included PAL and was a low-burden, highly sensitive, precise measure of cognitive function. The PALFAMS is the number of times a participant chose the correct box on their first attempt when recalling the pattern locations, calculated across all assessed trials. A higher number of events of selecting correct boxes indicates better cognitive function. Here, baseline was the last non-missing value prior to administration of the first dose of study intervention.
Time Frame: Baseline, Cycle 5 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, and Cycle 17 Day 1 (21 days cycle)
Population: The FAS included all the participants who were enrolled in the study and received at least 1 dose of treatment. The "number analyzed" refers to the number of participants included in the analysis at specific time points in each row.
Measure: Mean (Standard Deviation); unit: Number of Events
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 206 | 238
Number of Events
  Paired Assistance Learning (PAL) first attempt Memory score: Baseline | 10.9 (4.63) | 10.4 (4.71)
  PAL first attempt Memory score: Cycle 5 Day 1: number analyzed (Participants) | 163 | 195
  PAL first attempt Memory score: Cycle 5 Day 1 | 11.7 (4.81) | 10.8 (4.48)
  PAL first attempt Memory score: Cycle 9 Day 1: number analyzed (Participants) | 160 | 173
  PAL first attempt Memory score: Cycle 9 Day 1 | 12.5 (4.36) | 11.4 (4.59)
  PAL first attempt Memory score: Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  PAL first attempt Memory score: Cycle 13 Day 1 | 12.4 (4.86) | 11.8 (4.56)
  PAL first attempt Memory score: Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  PAL first attempt Memory score: Cycle 17 Day 1 | 13.2 (4.61) | 12.2 (5.07)

19. Secondary Outcome: Cognitive Functions Tests: Paired Associates Learning Total Errors Adjusted (PALTEA)
Description: The PAL is a computerized, self-completed cognitive test used to capture cognitive function, including attention, memory, and executive function. This gamified test included PALTEA and was a low-burden, highly sensitive, precise measure of cognitive function. PALTEA is the number of times a participant chose the incorrect box for a stimulus on assessment problems, plus an adjustment for the estimated number of errors they would have made on any problems, attempts, and recalls they did not reach. A higher number of events of selecting incorrect boxes indicates worse cognitive function. Here, baseline was the last non-missing value prior to administration of the first dose of study intervention.
Time Frame: Baseline, Cycle 5 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, and Cycle 17 Day 1 (21 days cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Number of Events
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 206 | 238
Number of Events
  PAL Total Errors (Adjusted): Baseline | 21.8 (17.18) | 24.8 (17.59)
  PAL Total Errors (Adjusted): Cycle 5 Day 1: number analyzed (Participants) | 163 | 195
  PAL Total Errors (Adjusted): Cycle 5 Day 1 | 19.2 (16.47) | 23.1 (17.53)
  PAL Total Errors (Adjusted): Cycle 9 Day 1: number analyzed (Participants) | 160 | 173
  PAL Total Errors (Adjusted): Cycle 9 Day 1 | 17.2 (15.17) | 21.5 (17.32)
  PAL Total Errors (Adjusted): Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  PAL Total Errors (Adjusted): Cycle 13 Day 1 | 17.5 (16.33) | 19.2 (16.31)
  PAL Total Errors (Adjusted): Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  PAL Total Errors (Adjusted): Cycle 17 Day 1 | 15.0 (14.92) | 19.2 (17.66)

20. Secondary Outcome: Cognitive Functions Tests: Reaction Time (RTI)
Description: This is a computerized, self-completed cognitive test used to capture cognitive function, including attention, memory, and executive function. This gamified test included Reaction Time Task (RTI) and was low-burden, highly sensitive, precise measures of cognitive function. RTI Median Five-Choice Movement Time: median time taken for a participant to release response button and select target stimulus after it flashed yellow on screen. Calculated across correct, assessed trials in which stimulus could appear in any one of five locations. RTI Median Five-Choice Reaction Time: median duration it took for a participant to release response button after presentation of target stimulus. Calculated across correct, assessed trials in which stimulus could appear in any one of five locations. Measured in milliseconds. Higher reaction times indicate worse cognitive function. Here, baseline was the last non-missing value prior to administration of the first dose of study intervention.
Time Frame: Baseline, Cycle 5 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, and Cycle 17 Day 1 (21 days cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 206 | 239
Millisecond (msec)
  Reaction time (RTI) Median Five-Choice Movement Time: Baseline | 314.7 (117.03) | 329.4 (141.24)
  RTI Median Five-Choice Movement Time: Cycle 5 Day 1: number analyzed (Participants) | 165 | 192
  RTI Median Five-Choice Movement Time: Cycle 5 Day 1 | 309.1 (94.85) | 310.5 (110.94)
  RTI Median Five-Choice Movement Time: Cycle 9 Day 1: number analyzed (Participants) | 160 | 170
  RTI Median Five-Choice Movement Time: Cycle 9 Day 1 | 305.3 (93.47) | 326.7 (106.02)
  RTI Median Five-Choice Movement Time: Cycle 13 Day 1: number analyzed (Participants) | 132 | 146
  RTI Median Five-Choice Movement Time: Cycle 13 Day 1 | 308.4 (89.55) | 324.1 (115.24)
  RTI Median Five-Choice Movement Time: Cycle 17 Day 1: number analyzed (Participants) | 94 | 113
  RTI Median Five-Choice Movement Time: Cycle 17 Day 1 | 319.6 (151.42) | 316.4 (96.69)
  RTI Median Five-Choice Reaction Time: Baseline | 401.3 (70.63) | 423.6 (115.56)
  RTI Median Five-Choice Reaction Time: Cycle 5 Day 1: number analyzed (Participants) | 165 | 192
  RTI Median Five-Choice Reaction Time: Cycle 5 Day 1 | 408.7 (119.26) | 413.0 (84.25)
  RTI Median Five-Choice Reaction Time: Cycle 9 Day 1: number analyzed (Participants) | 160 | 170
  RTI Median Five-Choice Reaction Time: Cycle 9 Day 1 | 401.5 (73.18) | 414.5 (67.68)
  RTI Median Five-Choice Reaction Time: Cycle 13 Day 1: number analyzed (Participants) | 132 | 146
  RTI Median Five-Choice Reaction Time: Cycle 13 Day 1 | 401.0 (63.56) | 412.3 (77.07)
  RTI Median Five-Choice Reaction Time: Cycle 17 Day 1: number analyzed (Participants) | 94 | 113
  RTI Median Five-Choice Reaction Time: Cycle 17 Day 1 | 396.8 (81.63) | 402.8 (51.93)

21. Secondary Outcome: Cognitive Functions Tests: Spatial Working Memory (SWM)
Description: The SWM is a computerized cognitive test. The SWM Between Errors (SWMBE) is number of times a participant incorrectly revisits a box in which a token has previously been found, calculated across all 4, 6, and 8 token trials. SWM Between Errors 4 Boxes (SWMBE4), SWM Between Errors 6 Boxes (SWMBE6), and SWM Between Errors 8 Boxes (SWMBE8) are number of times a participant revisits a box in which a token has previously been found. These are calculated across all trials with 4 tokens only for SWMBE4, 6 tokens only for SWMBE6, and 8 tokens only for SWMBE8. SWM Total Errors is number of times a box is selected that is certain not to contain a token and therefore should not have been visited by participant. A higher number of incorrect revisit events to previously found token boxes indicates worse cognitive function, and a lower number of revisit events indicates better cognitive function. Here, baseline was last non-missing value prior to administration of first dose of study intervention.
Time Frame: Baseline, Cycle 5 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, and Cycle 17 Day 1 (21 days cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Number of Events
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 206 | 237
Number of Events
  Spatial working memory (SWM) Between Errors: Baseline | 17.2 (8.89) | 18.6 (8.69)
  SWM Between Errors: Cycle 5 Day 1: number analyzed (Participants) | 162 | 192
  SWM Between Errors: Cycle 5 Day 1 | 15.5 (10.11) | 16.8 (8.39)
  SWM Between Errors: Cycle 9 Day 1: number analyzed (Participants) | 161 | 172
  SWM Between Errors: Cycle 9 Day 1 | 15.1 (9.78) | 16.3 (9.22)
  SWM Between Errors: Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  SWM Between Errors: Cycle 13 Day 1 | 13.4 (9.56) | 15.0 (8.85)
  SWM Between Errors: Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  SWM Between Errors: Cycle 17 Day 1 | 13.5 (9.48) | 13.7 (9.50)
  SWM Between Errors 4 Boxes: Baseline | 1.4 (1.39) | 1.4 (1.46)
  SWM Between Errors 4 Boxes: Cycle 5 Day 1: number analyzed (Participants) | 162 | 192
  SWM Between Errors 4 Boxes: Cycle 5 Day 1 | 1.0 (1.39) | 1.1 (1.42)
  SWM Between Errors 4 Boxes: Cycle 9 Day 1: number analyzed (Participants) | 161 | 172
  SWM Between Errors 4 Boxes: Cycle 9 Day 1 | 0.9 (1.33) | 1.1 (1.42)
  SWM Between Errors 4 Boxes: Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  SWM Between Errors 4 Boxes: Cycle 13 Day 1 | 0.8 (1.23) | 0.9 (1.37)
  SWM Between Errors 4 Boxes: Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  SWM Between Errors 4 Boxes: Cycle 17 Day 1 | 0.9 (1.32) | 0.7 (1.17)
  SWM Between Errors 6 Boxes: Baseline | 5.0 (3.44) | 5.2 (3.53)
  SWM Between Errors 6 Boxes: Cycle 5 Day 1: number analyzed (Participants) | 162 | 192
  SWM Between Errors 6 Boxes: Cycle 5 Day 1 | 4.3 (3.41) | 4.6 (3.42)
  SWM Between Errors 6 Boxes: Cycle 9 Day 1: number analyzed (Participants) | 161 | 172
  SWM Between Errors 6 Boxes: Cycle 9 Day 1 | 4.2 (3.64) | 4.7 (3.84)
  SWM Between Errors 6 Boxes: Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  SWM Between Errors 6 Boxes: Cycle 13 Day 1 | 3.2 (3.38) | 4.1 (3.34)
  SWM Between Errors 6 Boxes: Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  SWM Between Errors 6 Boxes: Cycle 17 Day 1 | 3.7 (3.25) | 4.0 (3.51)
  SWM Between Errors 8 Boxes: Baseline | 10.9 (5.66) | 12.1 (5.45)
  SWM Between Errors 8 Boxes: Cycle 5 Day 1: number analyzed (Participants) | 162 | 192
  SWM Between Errors 8 Boxes: Cycle 5 Day 1 | 10.2 (6.61) | 11.2 (5.31)
  SWM Between Errors 8 Boxes: Cycle 9 Day 1: number analyzed (Participants) | 161 | 172
  SWM Between Errors 8 Boxes: Cycle 9 Day 1 | 10.0 (6.31) | 10.5 (5.52)
  SWM Between Errors 8 Boxes: Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  SWM Between Errors 8 Boxes: Cycle 13 Day 1 | 9.3 (6.27) | 9.9 (5.91)
  SWM Between Errors 8 Boxes: Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  SWM Between Errors 8 Boxes: Cycle 17 Day 1 | 8.9 (6.42) | 9.0 (6.33)
  SWM Total Errors: Baseline | 17.5 (8.96) | 19.0 (8.75)
  SWM Total Errors: Cycle 5 Day 1: number analyzed (Participants) | 162 | 192
  SWM Total Errors: Cycle 5 Day 1 | 15.9 (10.24) | 17.3 (8.59)
  SWM Total Errors: Cycle 9 Day 1: number analyzed (Participants) | 161 | 172
  SWM Total Errors: Cycle 9 Day 1 | 15.5 (9.89) | 16.7 (9.42)
  SWM Total Errors: Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  SWM Total Errors: Cycle 13 Day 1 | 13.7 (9.71) | 15.3 (8.91)
  SWM Total Errors: Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  SWM Total Errors: Cycle 17 Day 1 | 13.8 (9.63) | 13.9 (9.63)

22. Secondary Outcome: Cognitive Functions Tests: Spatial Working Memory Strategy (SWMS)
Description: The SWM is a computerized cognitive test. The SWMS, the number of times a participant restarted search patterns from the same initial box, indicating their use of a planned strategy to find tokens. An increased number of events where search patterns started from the same initial box suggested participants were using a planned strategy to find tokens, which indicated better cognitive function. Here, a low score indicated high strategy use (1 = they always began the search from the same box). Conversely, high scores represented a decrease in events of beginning searches from the same box. Instead, starting from many different boxes suggested the participant was not using a consistent strategy, which indicated worse cognitive function. This was calculated across assessed trials with 6 tokens or more. Here, baseline was the last non-missing value prior to administration of the first dose of study intervention.
Time Frame: Baseline, Cycle 5 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, and Cycle 17 Day 1 (21 days cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Number of Events
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 206 | 237
Number of Events
  SWM Strategy (6-8 Boxes): Baseline | 8.8 (2.30) | 9.1 (2.32)
  SWM Strategy (6-8 Boxes): Cycle 5 Day 1: number analyzed (Participants) | 162 | 192
  SWM Strategy (6-8 Boxes): Cycle 5 Day 1 | 8.4 (2.80) | 8.8 (2.42)
  SWM Strategy (6-8 Boxes): Cycle 9 Day 1: number analyzed (Participants) | 161 | 172
  SWM Strategy (6-8 Boxes): Cycle 9 Day 1 | 8.2 (2.70) | 8.5 (2.44)
  SWM Strategy (6-8 Boxes): Cycle 13 Day 1: number analyzed (Participants) | 132 | 148
  SWM Strategy (6-8 Boxes): Cycle 13 Day 1 | 7.9 (3.18) | 8.6 (2.79)
  SWM Strategy (6-8 Boxes): Cycle 17 Day 1: number analyzed (Participants) | 93 | 114
  SWM Strategy (6-8 Boxes): Cycle 17 Day 1 | 7.9 (3.13) | 8.0 (3.08)

23. Secondary Outcome: St. George's Respiratory Questionnaire - Idiopathic (SGRQ-I) Pulmonary Fibrosis Version in Participants With Interstitial Lung Disease (ILD)/Pneumonitis
Description: The effect of T-DXd on symptoms, functioning, and HRQoL in HER2+ MBC participants with or without baseline brain metastasis was evaluated. The SGRQ-I is an idiopathic pulmonary fibrosis-specific version of the instrument developed and validated for use among participants with idiopathic pulmonary fibrosis, a type of ILD. The SGRQ-I was used to assess the HRQoL among participants who have been diagnosed with ILD/pneumonitis. It includes 34 of the original SGRQ items determined to be most reliable for assessing the HRQoL of participants with idiopathic pulmonary fibrosis. The instrument yields 3 domain scores (symptoms, activity, and impact) as well as a total score, with scores ranging from 0 to 100. Higher scores indicate greater impairment in HRQoL.
Time Frame: From time of ILD/pneumonitis diagnosis (every week) until end of safety follow-up (47 days post last dose) (up to 2 years 7 months)
Population: The safety analysis set- ILD consisted of participants who developed ILD/Pneumonitis. The "number analyzed" refers to the number of participants included in the analysis at specific time points in each row.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 14 | 27
Score on scale
  Total: Baseline | 32.1 (19.31) | 27.6 (20.97)
  Total: Week 1: number analyzed (Participants) | 4 | 7
  Total: Week 1 | 28.2 (17.10) | 33.1 (30.33)
  Total: Week 2: number analyzed (Participants) | 4 | 9
  Total: Week 2 | 23.3 (22.91) | 21.5 (14.48)
  Total: Week 3: number analyzed (Participants) | 4 | 8
  Total: Week 3 | 19.5 (20.10) | 15.3 (15.23)
  Total: Week 4: number analyzed (Participants) | 2 | 9
  Total: Week 4 | 4.2 (1.09) | 17.8 (15.49)
  Total: Week 5: number analyzed (Participants) | 2 | 9
  Total: Week 5 | 8.0 (6.40) | 15.9 (15.43)
  Total: Week 6: number analyzed (Participants) | 2 | 11
  Total: Week 6 | 6.7 (2.39) | 16.4 (11.95)
  Total: Week 7: number analyzed (Participants) | 3 | 9
  Total: Week 7 | 5.4 (3.49) | 14.8 (15.73)
  Total: Week 8: number analyzed (Participants) | 3 | 8
  Total: Week 8 | 3.3 (1.75) | 16.9 (17.04)
  Total: Week 9: number analyzed (Participants) | 2 | 8
  Total: Week 9 | 8.0 (4.29) | 23.3 (17.20)
  Total: Week 10: number analyzed (Participants) | 2 | 5
  Total: Week 10 | 6.6 (2.36) | 18.6 (14.54)
  Total: Week 11: number analyzed (Participants) | 2 | 6
  Total: Week 11 | 8.9 (1.79) | 20.3 (14.92)
  Total: Week 12: number analyzed (Participants) | 2 | 8
  Total: Week 12 | 8.4 (2.73) | 21.8 (14.40)
  Total: Week 13: number analyzed (Participants) | 2 | 6
  Total: Week 13 | 6.2 (0.27) | 20.4 (17.95)
  Total: Week 14: number analyzed (Participants) | 2 | 4
  Total: Week 14 | 5.5 (2.97) | 8.6 (7.19)
  Total: Week 15: number analyzed (Participants) | 2 | 6
  Total: Week 15 | 4.2 (1.09) | 12.9 (10.49)
  Total: Week 16: number analyzed (Participants) | 2 | 4
  Total: Week 16 | 4.2 (1.09) | 12.3 (10.10)
  Total: Week 17: number analyzed (Participants) | 2 | 4
  Total: Week 17 | 4.2 (1.09) | 12.1 (15.07)
  Total: Week 18: number analyzed (Participants) | 2 | 4
  Total: Week 18 | 4.2 (1.09) | 13.3 (16.29)
  Total: Week 19: number analyzed (Participants) | 3 | 3
  Total: Week 19 | 9.1 (7.02) | 8.7 (9.07)
  Total: Week 20: number analyzed (Participants) | 3 | 2
  Total: Week 20 | 7.9 (6.41) | 6.2 (3.86)
  Total: Week 21: number analyzed (Participants) | 3 | 4
  Total: Week 21 | 7.5 (5.78) | 5.2 (2.58)
  Total: Week 22: number analyzed (Participants) | 2 | 6
  Total: Week 22 | 6.7 (2.44) | 15.4 (13.24)
  Total: Week 23: number analyzed (Participants) | 2 | 5
  Total: Week 23 | 6.7 (2.44) | 9.8 (9.74)
  Total: Week 24: number analyzed (Participants) | 2 | 6
  Total: Week 24 | 6.7 (2.44) | 17.3 (15.09)
  Total: Week 25: number analyzed (Participants) | 3 | 5
  Total: Week 25 | 5.6 (2.56) | 11.0 (10.90)
  Total: Week 26: number analyzed (Participants) | 3 | 4
  Total: Week 26 | 5.6 (2.56) | 10.5 (10.81)
  Total: Week 27: number analyzed (Participants) | 3 | 5
  Total: Week 27 | 5.6 (2.56) | 13.5 (11.53)
  Total: Week 28: number analyzed (Participants) | 3 | 4
  Total: Week 28 | 5.6 (2.56) | 10.7 (11.13)
  Total: Week 29: number analyzed (Participants) | 2 | 5
  Total: Week 29 | 6.7 (2.44) | 16.5 (16.52)
  Total: Week 30: number analyzed (Participants) | 3 | 6
  Total: Week 30 | 4.7 (1.19) | 19.6 (18.60)
  Total: Week 31: number analyzed (Participants) | 3 | 5
  Total: Week 31 | 5.6 (2.56) | 15.9 (13.98)
  Total: Week 32: number analyzed (Participants) | 3 | 4
  Total: Week 32 | 5.6 (2.56) | 11.4 (10.89)
  Total: Week 33: number analyzed (Participants) | 2 | 3
  Total: Week 33 | 6.7 (2.44) | 5.2 (3.15)
  Total: Week 34: number analyzed (Participants) | 3 | 3
  Total: Week 34 | 5.5 (2.62) | 11.9 (10.36)
  Total: Week 35: number analyzed (Participants) | 3 | 3
  Total: Week 35 | 6.6 (2.76) | 11.9 (10.32)
  Total: Week 36: number analyzed (Participants) | 2 | 2
  Total: Week 36 | 6.7 (2.44) | 15.9 (17.62)
  Total: Week 37: number analyzed (Participants) | 4 | 3
  Total: Week 37 | 5.4 (2.45) | 11.5 (9.72)
  Total: Week 38: number analyzed (Participants) | 2 | 3
  Total: Week 38 | 6.7 (2.44) | 11.8 (10.13)
  Total: Week 39: number analyzed (Participants) | 1 | 2
  Total: Week 39 | 5.0 (NA) — Since the number of participants is 1, SD was not calculable. | 6.2 (3.86)
  Total: Week 40: number analyzed (Participants) | 3 | 2
  Total: Week 40 | 5.6 (2.56) | 6.2 (3.86)
  Total: Week 41: number analyzed (Participants) | 3 | 1
  Total: Week 41 | 5.6 (2.56) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 42: number analyzed (Participants) | 2 | 2
  Total: Week 42 | 6.7 (2.44) | 6.2 (3.86)
  Total: Week 43: number analyzed (Participants) | 3 | 2
  Total: Week 43 | 5.6 (2.56) | 6.2 (3.86)
  Total: Week 44: number analyzed (Participants) | 3 | 2
  Total: Week 44 | 7.4 (5.54) | 6.2 (3.86)
  Total: Week 45: number analyzed (Participants) | 1 | 2
  Total: Week 45 | 9.5 (NA) — Since the number of participants is 1, SD was not calculable. | 6.2 (3.86)
  Total: Week 46: number analyzed (Participants) | 2 | 1
  Total: Week 46 | 6.7 (2.44) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 47: number analyzed (Participants) | 2 | 2
  Total: Week 47 | 6.7 (2.44) | 6.2 (3.86)
  Total: Week 48: number analyzed (Participants) | 2 | 2
  Total: Week 48 | 6.7 (2.44) | 6.2 (3.86)
  Total: Week 49: number analyzed (Participants) | 2 | 1
  Total: Week 49 | 6.7 (2.44) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 50: number analyzed (Participants) | 2 | 2
  Total: Week 50 | 9.1 (0.99) | 6.2 (3.86)
  Total: Week 51: number analyzed (Participants) | 2 | 1
  Total: Week 51 | 8.2 (0.32) | 10.4 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 52: number analyzed (Participants) | 2 | 0
  Total: Week 52 | 6.7 (2.44) |
  Total: Week 53: number analyzed (Participants) | 2 | 1
  Total: Week 53 | 6.7 (2.44) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 54: number analyzed (Participants) | 2 | 1
  Total: Week 54 | 6.7 (2.44) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 55: number analyzed (Participants) | 2 | 1
  Total: Week 55 | 6.7 (2.44) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 56: number analyzed (Participants) | 2 | 1
  Total: Week 56 | 7.5 (3.53) | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 57: number analyzed (Participants) | 1 | 1
  Total: Week 57 | 8.4 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 58: number analyzed (Participants) | 1 | 1
  Total: Week 58 | 8.4 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 59: number analyzed (Participants) | 1 | 1
  Total: Week 59 | 10.0 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 60: number analyzed (Participants) | 1 | 1
  Total: Week 60 | 8.4 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 61: number analyzed (Participants) | 1 | 1
  Total: Week 61 | 8.4 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 62: number analyzed (Participants) | 1 | 1
  Total: Week 62 | 8.4 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 63: number analyzed (Participants) | 1 | 1
  Total: Week 63 | 10.0 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 64: number analyzed (Participants) | 1 | 1
  Total: Week 64 | 8.4 (NA) — Since the number of participants is 1, SD was not calculable. | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 65: number analyzed (Participants) | 0 | 1
  Total: Week 65 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 66: number analyzed (Participants) | 0 | 1
  Total: Week 66 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 67: number analyzed (Participants) | 0 | 1
  Total: Week 67 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 68: number analyzed (Participants) | 0 | 1
  Total: Week 68 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 69: number analyzed (Participants) | 0 | 1
  Total: Week 69 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 70: number analyzed (Participants) | 0 | 1
  Total: Week 70 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 71: number analyzed (Participants) | 0 | 1
  Total: Week 71 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  Total: Week 72: number analyzed (Participants) | 0 | 1
  Total: Week 72 |  | 8.9 (NA) — Since the number of participants is 1, SD was not calculable.
  End of treatment: number analyzed (Participants) | 4 | 9
  End of treatment | 31.1 (18.65) | 18.0 (19.16)
  Safety Follow-up: number analyzed (Participants) | 2 | 2
  Safety Follow-up | 23.4 (6.38) | 21.4 (25.36)

24. Secondary Outcome: MD Anderson Symptom Inventory Brain Tumor-Specific Items in Brain Metastasis at Baseline Participants
Description: The T-DXd on symptoms, functioning, and HRQoL in HER2+ MBC participants with or without baseline brain metastasis was evaluated. The MDASI brain tumor module includes 9 symptoms specific to brain tumors (weakness on one side of the body, difficulty understanding, difficulty speaking, seizures, difficulty concentrating, problems with vision, change in appearance, change in bowel pattern (diarrhea or constipation), and irritability). These 9 items will be used to capture symptoms associated with brain metastasis for those diagnosed with brain metastasis. Each item is rated on an 11-point numeric rating scale on a scale of 0-10, with higher scores indicating greater symptom severity. Here, baseline was the last non-missing value prior to administration of the first dose of study intervention.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, and Cycle 39 Day 1 (21 days cycle)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 213
Score on scale
  Change in Appearance at Its Worst: Baseline | 1.8 (2.44)
  Change in Appearance at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Change in Appearance at Its Worst: Cycle 2 Day 1 | 1.9 (2.44)
  Change in Appearance at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 170
  Change in Appearance at Its Worst: Cycle 3 Day 1 | 2.1 (2.51)
  Change in Appearance at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Change in Appearance at Its Worst: Cycle 4 Day 1 | 1.9 (2.20)
  Change in Appearance at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 166
  Change in Appearance at Its Worst: Cycle 5 Day 1 | 2.1 (2.45)
  Change in Appearance at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Change in Appearance at Its Worst: Cycle 39 Day 1 | 3.0 (NA) — Since there is only 1 participant, SD was not calculable.
  Change in Bowel Pattern at Its Worst: Baseline | 1.7 (2.46)
  Change in Bowel Pattern at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Change in Bowel Pattern at Its Worst: Cycle 2 Day 1 | 2.5 (2.55)
  Change in Bowel Pattern at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 170
  Change in Bowel Pattern at Its Worst: Cycle 3 Day 1 | 2.7 (2.67)
  Change in Bowel Pattern at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Change in Bowel Pattern at Its Worst: Cycle 4 Day 1 | 3.0 (2.74)
  Change in Bowel Pattern at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 166
  Change in Bowel Pattern at Its Worst: Cycle 5 Day 1 | 2.8 (2.69)
  Change in Bowel Pattern at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Change in Bowel Pattern at Its Worst: Cycle 39 Day 1 | 0 (NA) — Since there is only 1 participant, SD was not calculable.
  Difficulty Concentrating at Its Worst: Baseline | 1.8 (2.23)
  Difficulty Concentrating at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Difficulty Concentrating at Its Worst: Cycle 2 Day 1 | 1.7 (2.03)
  Difficulty Concentrating at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 170
  Difficulty Concentrating at Its Worst: Cycle 3 Day 1 | 1.9 (2.27)
  Difficulty Concentrating at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Difficulty Concentrating at Its Worst: Cycle 4 Day 1 | 1.6 (2.03)
  Difficulty Concentrating at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 165
  Difficulty Concentrating at Its Worst: Cycle 5 Day 1 | 1.5 (1.95)
  Difficulty Concentrating at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Difficulty Concentrating at Its Worst: Cycle 39 Day 1 | 1.0 (NA) — Since there is only 1 participant, SD was not calculable.
  Difficulty Speaking at Its Worst: Baseline | 1.4 (2.18)
  Difficulty Speaking at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Difficulty Speaking at Its Worst: Cycle 2 Day 1 | 1.3 (1.96)
  Difficulty Speaking at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 169
  Difficulty Speaking at Its Worst: Cycle 3 Day 1 | 1.4 (1.97)
  Difficulty Speaking at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 161
  Difficulty Speaking at Its Worst: Cycle 4 Day 1 | 1.1 (1.80)
  Difficulty Speaking at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 166
  Difficulty Speaking at Its Worst: Cycle 5 Day 1 | 1.3 (1.98)
  Difficulty Speaking at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Difficulty Speaking at Its Worst: Cycle 39 Day 1 | 1.0 (NA) — Since there is only 1 participant, SD was not calculable.
  Difficulty Understanding at Its Worst: Baseline | 1.5 (2.29)
  Difficulty Understanding at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Difficulty Understanding at Its Worst: Cycle 2 Day 1 | 0.9 (1.67)
  Difficulty Understanding at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 169
  Difficulty Understanding at Its Worst: Cycle 3 Day 1 | 1.2 (1.87)
  Difficulty Understanding at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Difficulty Understanding at Its Worst: Cycle 4 Day 1 | 1.0 (1.83)
  Difficulty Understanding at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 166
  Difficulty Understanding at Its Worst: Cycle 5 Day 1 | 0.9 (1.68)
  Difficulty Understanding at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Difficulty Understanding at Its Worst: Cycle 39 Day 1 | 0 (NA) — Since there is only 1 participant, SD was not calculable.
  Irritability at its Worst: Baseline | 1.8 (2.27)
  Irritability at its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Irritability at its Worst: Cycle 2 Day 1 | 1.9 (2.23)
  Irritability at its Worst: Cycle 3 Day 1: number analyzed (Participants) | 169
  Irritability at its Worst: Cycle 3 Day 1 | 1.8 (2.04)
  Irritability at its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Irritability at its Worst: Cycle 4 Day 1 | 1.9 (2.06)
  Irritability at its Worst: Cycle 5 Day 1: number analyzed (Participants) | 166
  Irritability at its Worst: Cycle 5 Day 1 | 1.9 (2.12)
  Irritability at its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Irritability at its Worst: Cycle 39 Day 1 | 4.0 (NA) — Since there is only 1 participant, SD was not calculable.
  Seizures at Its Worst: Baseline | 0.5 (1.58)
  Seizures at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Seizures at Its Worst: Cycle 2 Day 1 | 0.5 (1.38)
  Seizures at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 170
  Seizures at Its Worst: Cycle 3 Day 1 | 0.5 (1.52)
  Seizures at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Seizures at Its Worst: Cycle 4 Day 1 | 0.5 (1.47)
  Seizures at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 165
  Seizures at Its Worst: Cycle 5 Day 1 | 0.5 (1.40)
  Seizures at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Seizures at Its Worst: Cycle 39 Day 1 | 0 (NA) — Since there is only 1 participant, SD was not calculable.
  Vision at Its Worst: Baseline | 1.6 (2.28)
  Vision at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Vision at Its Worst: Cycle 2 Day 1 | 1.6 (2.24)
  Vision at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 169
  Vision at Its Worst: Cycle 3 Day 1 | 1.5 (2.10)
  Vision at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 162
  Vision at Its Worst: Cycle 4 Day 1 | 1.4 (1.94)
  Vision at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 165
  Vision at Its Worst: Cycle 5 Day 1 | 1.5 (2.01)
  Vision at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Vision at Its Worst: Cycle 39 Day 1 | 1.0 (NA) — Since there is only 1 participant, SD was not calculable.
  Weakness on One Body Side at Its Worst: Baseline | 2.1 (2.54)
  Weakness on One Body Side at Its Worst: Cycle 2 Day 1: number analyzed (Participants) | 174
  Weakness on One Body Side at Its Worst: Cycle 2 Day 1 | 1.7 (2.35)
  Weakness on One Body Side at Its Worst: Cycle 3 Day 1: number analyzed (Participants) | 169
  Weakness on One Body Side at Its Worst: Cycle 3 Day 1 | 1.8 (2.28)
  Weakness on One Body Side at Its Worst: Cycle 4 Day 1: number analyzed (Participants) | 161
  Weakness on One Body Side at Its Worst: Cycle 4 Day 1 | 1.8 (2.48)
  Weakness on One Body Side at Its Worst: Cycle 5 Day 1: number analyzed (Participants) | 166
  Weakness on One Body Side at Its Worst: Cycle 5 Day 1 | 1.6 (2.18)
  Weakness on One Body Side at Its Worst: Cycle 39 Day 1: number analyzed (Participants) | 1
  Weakness on One Body Side at Its Worst: Cycle 39 Day 1 | 0 (NA) — Since there is only 1 participant, SD was not calculable.

25. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of the participants who received T-DXd was evaluated.
  SAE=Serious adverse events; CTCAE=Common Terminology for Adverse Events
Time Frame: From first dose until end of safety follow-up (47 days post last dose) (up to 2 years 7 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241 | 263
Participants
  Any AE | 237 | 259
  Any AE, excluding AEs associated with COVID-19 | 237 | 259
  Any AE associated with COVID-19 | 45 | 54
  Any AE possibly related to treatment | 230 | 242
  Any AE of CTCAE grade 3 or higher | 118 | 134
  Any AE of CTCAE grade 3 or higher, possibly related to treatment | 98 | 100
  Any AE with outcome = death | 6 | 8
  Any AE with outcome = death, excluding AEs associated with COVID-19 | 6 | 8
  Any AE with outcome = death, associated with COVID-19 | 0 | 0
  Any AE with outcome = death, possibly related to treatment | 5 | 6
  Any SAE (events with outcome = death) | 46 | 62
  Any SAE (events with outcome = death), possibly related to treatment | 25 | 25
  Any AE leading to dose reduction | 65 | 60
  Any AE leading to dose reduction, possibly related to treatment | 63 | 53
  Any AE leading to dose interruption | 124 | 146
  Any AE leading to dose interruption, possibly related to treatment | 82 | 83
  Any AE leading to discontinuation of treatment | 23 | 40
  Any AE leading to discontinuation of treatment, excluding AEs associated with COVID-19 | 23 | 39
  Any AE leading to discontinuation of treatment, associated with COVID-19 | 0 | 1
  Any AE leading to discontinuation of treatment, possibly related to treatment | 20 | 34
  Any SAE leading to discontinuation of treatment | 8 | 18
  Any SAE leading to discontinuation of treatment, possibly related to treatment | 6 | 13
  Any Other Adverse events (OAE) | 0 | 5
  Any Adverse event of special event | 54 | 71

26. Secondary Outcome: Number of Participants With Investigator-assessed ILD/Pneumonitis
Description: The number of participants with ILD/Pneumonitis were by grouped term based on Investigator-reported preferred terms. No adjudication was performed.
Time Frame: From first dose until end of safety follow-up (47 days post last dose) (up to 2 years 7 months)
Population: The Safety analysis set consisted of all participants who had received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 241 | 263
Participants
  Interstitial lung disease | 19 | 17
  Lung opacity | 2 | 0
  Pneumonitis | 10 | 24
  Pulmonary fibrosis | 1 | 1
  Radiation pneumonitis | 1 | 0
  Lung infiltration | 0 | 1

27. Secondary Outcome: Number of Participants With ILD Clinical Symptoms Resolution Among ILD/Pneumonitis Participants Who Have Been Treated With High Dose Steroid
Description: The number of participants with ILD clinical symptoms resolution in ILD/Pneumonitis participants who have been treated with high dose steroid (>2 mg dexamethasone) were evaluated.
Time Frame: From first dose until end of safety follow-up (47 days post last dose) (up to 2 years 7 months)
Population: The Safety analysis set-ILD consisted of all participants who had developed ILD/Pneumonitis. Here, the "overall number of participants analyzed" represents those who were treated with a high dose of steroids. Participants could have multiple ILD events with different statuses.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
Number analyzed (Participants) | 26 | 39
Participants
  Resolved: Recovered/resolved | 18 | 24
  Resolved: Recovering/resolving | 1 | 2
  Resolved: Recovered/resolved with sequelae | 1 | 1
  Unresolved: Not recovered/resolved | 6 | 6
  Unresolved: Fatal | 3 | 6

ADVERSE EVENTS:
Time Frame: From first dose until end of safety follow-up (47 days post last dose) (up to 2 years 7 months)
Arm/Group | Cohort 1: Trastuzumab Deruxtecan (T-DXd) | Cohort 2: Trastuzumab Deruxtecan (T-DXd)
All-Cause Mortality (participants affected / at risk) | 41/241 | 43/263
Serious Adverse Events (participants affected / at risk) | 46/241 | 62/263
Other Adverse Events (participants affected / at risk) | 235/241 | 253/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Trastuzumab Deruxtecan (T-DXd) (N=241) | Cohort 2: Trastuzumab Deruxtecan (T-DXd) (N=263)
Campylobacter colitis (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 3
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 0 | 2
Citrobacter sepsis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 4
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Hemianopia homonymous (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 5
Cardiac tamponade (Cardiac disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 6
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Pseudocirrhosis (Hepatobiliary disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 2
Gait disturbance (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Trastuzumab Deruxtecan (T-DXd) (N=241) | Cohort 2: Trastuzumab Deruxtecan (T-DXd) (N=263)
COVID-19 (Infections and infestations) | 40 | 50
Nasopharyngitis (Infections and infestations) | 17 | 26
Upper respiratory tract infection (Infections and infestations) | 15 | 19
Urinary tract infection (Infections and infestations) | 21 | 29
Anaemia (Blood and lymphatic system disorders) | 62 | 67
Leukopenia (Blood and lymphatic system disorders) | 15 | 15
Neutropenia (Blood and lymphatic system disorders) | 63 | 58
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 23
Decreased appetite (Metabolism and nutrition disorders) | 44 | 54
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 16
Insomnia (Psychiatric disorders) | 21 | 28
Dizziness (Nervous system disorders) | 17 | 23
Dysgeusia (Nervous system disorders) | 22 | 0
Headache (Nervous system disorders) | 48 | 55
Paraesthesia (Nervous system disorders) | 16 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 22
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 17 | 14
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Abdominal pain (Gastrointestinal disorders) | 18 | 17
Abdominal pain upper (Gastrointestinal disorders) | 32 | 26
Constipation (Gastrointestinal disorders) | 98 | 105
Diarrhoea (Gastrointestinal disorders) | 85 | 74
Dyspepsia (Gastrointestinal disorders) | 33 | 22
Nausea (Gastrointestinal disorders) | 171 | 168
Stomatitis (Gastrointestinal disorders) | 32 | 24
Vomiting (Gastrointestinal disorders) | 80 | 73
Alopecia (Skin and subcutaneous tissue disorders) | 83 | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 0
Asthenia (General disorders) | 103 | 71
Fatigue (General disorders) | 77 | 95
Oedema peripheral (General disorders) | 19 | 14
Pyrexia (General disorders) | 35 | 30
Alanine aminotransferase increased (Investigations) | 26 | 36
Aspartate aminotransferase increased (Investigations) | 38 | 31
Blood bilirubin increased (Investigations) | 16 | 0
Ejection fraction decreased (Investigations) | 23 | 29
Gamma-glutamyl transferase increased (Investigations) | 18 | 16
Neutrophil count decreased (Investigations) | 27 | 24
Platelet count decreased (Investigations) | 16 | 16
Weight decreased (Investigations) | 0 | 19
White blood cell count decreased (Investigations) | 0 | 18
Dry eye (Eye disorders) | 0 | 19
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04739761/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04739761/SAP_001.pdf